CLINICAL TRIAL: NCT01461473
Title: R01: Comparative Outcomes Management With Electronic Data Technology (COMET) Study
Brief Title: Comparative Outcomes Management With Electronic Data Technology (COMET) Study
Acronym: COMET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Clete A. Kushida, Principal Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SU-10182011-8536; 1R01HS019738-01 (AHRQ)
Record Dates: First submitted 2011-10-20; First posted 2011-10-28 (Estimated); Results first posted 2017-05-17 (Actual); Last update posted 2017-05-17 (Actual); Status verified 2017-04

CONDITIONS: Sleep Apnea, Obstructive
Keywords: Obstructive Sleep Apnea; Obstructive Sleep Apnea Syndrome; Sleep Apnea Syndrome, Obstructive; Syndrome, Obstructive Sleep Apnea; Syndrome, Sleep Apnea, Obstructive; Syndrome, Upper Airway Resistance, Sleep Apnea; Upper Airway Resistance Sleep Apnea Syndrome
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Occlusal Splints

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Positive Airway Pressure (Active Comparator): Participants randomized to standard clinical Positive Airway Pressure (PAP) treatment for Obstructive Sleep Apnea (OSA).
  Interventions: Device: Positive Airway Pressure (PAP)
- Oral Appliance (Active Comparator): Subjects randomized to standard Oral Appliance (OA) treatment for Obstructive Sleep Apnea (OSA).
  Interventions: Device: Oral Appliance (OA)

INTERVENTIONS:
Device: Positive Airway Pressure (PAP) — Participants randomized to the Positive Airway Pressure treatment group received adequate Positive Airway Pressure (PAP) pressure therapy by a PAP titration study and used the device for 6 months.
  Other Names: Auto-titrating PAP (APAP), Continuous PAP (CPAP)
  Arms: Positive Airway Pressure
Device: Oral Appliance (OA) — Participants randomized to the Oral Appliance treatment group received a dental evaluation to determine the optimal setting for the Oral Appliance (OA), and used the appliance for 6 months.
  Other Names: Mandibular Advancement Device
  Arms: Oral Appliance

SUMMARY:
STAGE I of the COMET study was to develop an Electronic Network Informatics Infrastructure that prospectively enabled access to and the sharing of clinical and research data.

STAGE II: This was a Comparative Effectiveness Trial (CET) evaluating positive airway pressure (PAP) vs. oral appliance (OA) therapy in improving hypertension and abnormalities in cardiovascular function in overweight/obese patients with obstructive sleep apnea (OSA). Data collected during the STAGE II study was incorporated in Part 3 of the STAGE I study.

STAGE III of the COMET study was completion of data analysis and preparation of the electronic network informatics infrastructure for use beyond the four Clinical Centers to interested CTSA institutions. We also explored expanding ontologies, and the use of federated database methodology.

DETAILED DESCRIPTION:
STAGE I, Part 1: We extracted limited access data sets from an existing research database (prior research patients' data from APPLES research project, where patients consented to provide a limited access data sets to the public domain as required by grants funded by the National Heart, Lung, and Blood Institute [NHLBI], PI: Dr. Clete Kushida) and a dummy database with prepared test data (no real patient data) to evaluate and refine the initial iterations of the informatics infrastructure created via an agile evolutionary development process.

STAGE I, Part 2: We expanded the functionality of the informatics infrastructure by testing its ability to incorporate research data collected from an electronic questionnaire, the Alliance Sleep Questionnaire (ASQ). We enabled data collection using the ASQ in order to use these data to evaluate and refine the iterations for the informatics infrastructure.

STAGE I, Part 3: We expanded the functionality of the informatics infrastructure by testing its ability to incorporate live (ongoing) longitudinal data collected from multiple forms and data sources obtained during the STAGE II study. The addition of these data allowed the COMET Steering Committee to create use cases with a greater diversity of data content. The STAGE II data were used to evaluate and refine the iterations for the expanded informatics infrastructure.

STAGE I, Part 4: Part 4 was designed to expand the collection of data beyond individual research studies, tapping into University-wide systems (e.g., Stride) to link longitudinal data collected during research studies to longitudinal data collected during clinical visits. Only de-identified data were shared with the network, and only the local site held the codebook that translated the Global Identifier (ID) to the Participant ID. All Health Insurance Portability and Accountability Act (HIPAA) regulations were considered.

STAGE II: This stage was comprised of the multicenter, randomized, parallel group, comparative effectiveness trial to compare positive airway pressure (PAP) vs. oral appliance (OA) therapy in improving hypertension and abnormalities in cardiovascular function in overweight/obese patients with obstructive sleep apnea (OSA). Data collected during the STAGE II study were incorporated in Part 3 of the STAGE I study. This comparative effectiveness trial was conducted at 4 clinical centers, and the data collected during this trial were used to test the electronic network informatics infrastructure. The primary aim of the Stage II CET was to evaluate and compare the effect of positive airway pressure and oral appliance therapy on 24-hour blood pressure and vascular structure and function associated with obstructive sleep apnea in a primarily female, overweight/obese hypertensive population.

STAGE III: This stage was comprised of completion of data analysis and preparation of the electronic network informatics infrastructure for deployment beyond the four Clinical Centers to interested Clinical and Translational Science Awards (CTSA) institutions. We also explored expanding the ontologies beyond a sleep-related ontology to other medical ontologies, and the use of federated database methodology.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* BMI > = 25.0 kg/m^2.
* A diagnosis of obstructive sleep apnea based upon medical history and apnea- hypopnea index > = 10.0 or oxygen desaturation index (ODI; ≥4%) ≥ 10.0 on Diagnostic Polysomnogram.
* Report a history of hypertension (or need for treatment for hypertension) which is currently untreated OR taking medication for the treatment of hypertension.
* Stable medication regimen for 2 months prior to the Baseline Testing Visit. As-needed medications such as those used for allergy, cold, or minor pain symptoms may be used at the discretion of the Clinical Center physician.

Exclusion Criteria:

* Cardiovascular disease which, in the judgment of the investigator, if observed during standard clinical practice would lead the treating physician to make every effort to treat the patient's sleep apnea with positive airway pressure, rather than alternative treatments.
* Clinically significant acute or chronic disease that is not well controlled or could affect ability to complete or comply with study procedures, in the opinion of the Clinical Center physician.
* Respiratory disease requiring supplemental oxygen or medication. Individuals with asthma may be included at the discretion of the Clinical Center physician if disease is well controlled and medications are stable for 2 months.
* History of (within 12 months prior to enrollment), or current diagnosis of, Axis I or Axis II psychiatric disorder (other than obstructive sleep apnea) that in the opinion of the Clinical Center physician would affect ability to complete or comply with study procedures (e.g., schizophrenia and other psychotic disorders).
* History of (within 3 months prior to enrollment), or current diagnosis of narcolepsy, idiopathic hypersomnia, restless legs syndrome, rapid eye movement (REM) behavior disorder, persistent situational insomnia, or sleep-related breathing disorders other than obstructive sleep apnea.
* Periodic limb movement arousal index > 10.0 on the Diagnostic Polysomnogram.
* Significant daytime sleepiness at study entry as indicated by:

  * an Epworth Sleepiness Scale total score > 16, or a score of 3 (high chance) on the question about risk of dozing "In a car, while stopped for a few minutes in traffic" or
  * a report of falling asleep at the wheel, a motor vehicle accident, or near-miss accident due to sleepiness in the past 24 months, which in the judgment of the study physician was not attributable to acute sleep loss.
* Oxygen saturation < 80% for > 10% of sleep time during the Diagnostic Polysomnogram, or intervention with positive airway pressure or oxygen for safety purposes during the Diagnostic Polysomnogram.
* Any prior treatment for obstructive sleep apnea with positive airway pressure or oral appliance, or surgical treatment for obstructive sleep apnea in the past year.
* Contraindication for treatment with either positive airway pressure or oral appliance, in the opinion of the Clinical Center physician or dentist, including significant nasal obstruction, insufficient or loose teeth, dentures, advanced periodontal disease, or significant temporomandibular joint pain.
* Pregnancy.
* Difficulty understanding or speaking English, or inability to read and understand informed consent and study procedures.
* Significant vision, hearing, or motor problems that, in the opinion of the Clinical Center physician, would affect ability to complete study procedures.
* A work schedule that does not allow for nighttime sleep on the 3 nights before each study visit.
* Current or planned participation in another research study.
* Metal objects, devices, or implants that are in or on the body (Stanford Clinical Center only).
* Creatinine clearance <30 and creatinine >1.6 (Stanford Clinical Center only).
* Upper arm circumference > 20 inches

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2011-12; Primary Completion 2014-05 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clete A Kushida, MD, PhD, Study Director — Stanford University; Allan Pack, MD, Principal Investigator — Center for Sleep, University of Pennsylvania School of Medicine; Susan Redline, MD, Principal Investigator — Harvard Brigham and Women's Hospital; Ruth Benca, MD, Principal Investigator — University of Wisconsin-Madison School of Medicine
Locations (4):
- United States (4):
  - Stanford Sleep Medicine Center, Redwood City, California
  - Harvard Brigham and Women's Hospital, Boston, Massachusetts
  - Center for Sleep and Circadian Neurobiology, University of Pennsylvania School of Medicine, Philadelphia, Pennsylvania
  - University of Wisconsin-Madison School of Medicine, Department of Psychiatry, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Young T, Palta M, Dempsey J, Skatrud J, Weber S, Badr S. The occurrence of sleep-disordered breathing among middle-aged adults. N Engl J Med. 1993 Apr 29;328(17):1230-5. doi: 10.1056/NEJM199304293281704. PMID 8464434
- [Background] Nichols DA, DeSalvo S, Miller RA, Jonsson D, Griffin KS, Hyde PR, Walsh JK, Kushida CA. The COMET Sleep Research Platform. EGEMS (Wash DC). 2014 Nov 24;2(1):1059. doi: 10.13063/2327-9214.1059. eCollection 2014. PMID 25848590

RESULTS

PARTICIPANT FLOW:
Groups:
- Positive Airway Pressure: Participants randomized to standard clinical Positive Airway Pressure (PAP) treatment for Obstructive Sleep Apnea (OSA).
  Positive Airway Pressure: Participants who are randomized to the Positive Airway Pressure treatment group will receive adequate Positive Airway Pressure (PAP) pressure setting through standard clinical polysomnography (PSG) study.
- Oral Appliance: Subjects randomized to standard Oral Appliance (OA) treatment for Obstructive Sleep Apnea (OSA).
  Oral Appliance: Participants who are randomized to the Oral Appliance Treatment Group will receive a dental evaluation to determine the optimal setting for the Oral Appliance (OA) device.
Period: Overall Study
Arm/Group | Positive Airway Pressure | Oral Appliance
Started | 72 | 59
Completed | 67 | 55
Not Completed | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Positive Airway Pressure | Oral Appliance | Total
Number analyzed (Participants) | 72 | 59 | 131
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.85 (12.17) | 52.61 (9.84) | 53.84 (11.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 17 | 37
  Male | 52 | 42 | 94
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 6 | 9
  Not Hispanic or Latino | 69 | 53 | 122
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 5 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 4 | 8
  White | 62 | 49 | 111
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 72 | 59 | 131

OUTCOME MEASURES:

1. Primary Outcome: Nocturnal Mean Arterial Blood Pressure (NMAP) at 2 Months
Description: Mean arterial blood pressure during the sleep period as recorded by 24-hour ambulatory blood pressure monitoring after approximately 2 months of treatment
Time Frame: 2 months
Population: 31 participants in the Positive Airway Pressure arm and 29 participants in the Oral Appliance arm failed to return for 24-hour ambulatory blood pressure monitoring at the two-months time point, but did return at the six-month time point for blood pressure monitoring at the six-month time point and to complete the study.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Positive Airway Pressure | Oral Appliance
Number analyzed (Participants) | 36 | 26
mmHg | 82.1 (7.79) | 84.3 (9.60)
Statistical Analysis 1: Comparison: Positive Airway Pressure vs Oral Appliance; These data were analyzed using an analysis of covariance via general linear model (GLM). The GLM has an indicator variable for PAP vs. OA plus covariates for baseline apnea-hypopnea index, gender, site and baseline NMAP. The primary hypothesis tested is that the 2-month means differ between study arms, after adjustment for the above covariates. A Wald statistic was constructed for hypothesis testing; Test type: Superiority or Other; p = 0.2067, Analysis of covariance (GLM)

2. Secondary Outcome: Nocturnal Mean Arterial Blood Pressure (NMAP) at 6 Months
Description: Nocturnal mean arterial blood pressure as recorded by 24-hour ambulatory blood pressure monitoring after approximately 6 months of treatment
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Positive Airway Pressure | Oral Appliance
Number analyzed (Participants) | 67 | 55
mmHg | 83.1 (9.63) | 84.7 (9.59)
Statistical Analysis 1: Comparison: Positive Airway Pressure vs Oral Appliance; Generalized linear mixed model (GLMM) was fit in which the outcome was regressed on an indicator variable for PAP vs. OA, baseline apnea-hypopnea index, gender, site and baseline value of the outcome. A Wald statistic was constructed for hypothesis testing; Test type: Superiority or Other; p = 0.3902, GLMM

3. Secondary Outcome: Ratio of Nocturnal Mean Arterial Pressure (NMAP) to Daytime Mean Arterial Pressure at 2 Months
Description: Ratio of NMAP to mean daytime arterial pressure, expressed as a percentage at the 2 month visit for PAP and OA arms. The ratio is calculated by dividing the NMAP by the daytime mean arterial pressure; the result is then multiplied by 100 to obtain a percentage.
Time Frame: 2 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of NMAP to daytime MAP
Arm/Group | Positive Airway Pressure | Oral Appliance
Number analyzed (Participants) | 36 | 26
percentage of NMAP to daytime MAP | 86.8 (7.07) | 87.0 (7.67)
Statistical Analysis 1: Comparison: Positive Airway Pressure vs Oral Appliance; A GLMM was fit in which the outcome was regressed on an indicator variable for PAP vs. OA, baseline apnea-hypopnea index, gender, site and baseline value of the outcome. A Wald statistic was constructed for hypothesis testing; Test type: Superiority or Other; p = 0.9319, GLMM

4. Secondary Outcome: Ratio of NMAP to Daytime Mean Arterial Pressure at 6 Months
Description: Ratio of NMAP to daytime mean arterial pressure, expressed as a percentage at the 6 month visit for PAP and OA arms. The ratio is calculated by dividing the NMAP by the daytime mean arterial pressure; the result is then multiplied by 100 to obtain a percentage.
Time Frame: 6 months
Population: Two participants in the PAP arm and 1 participant in the OA arm did not have sufficient daytime MAP data to calculate the ratio of NMAP to daytime MAP at 6 months
Measure: Mean (Standard Deviation); unit: percentage of NMAP to daytime MAP
Arm/Group | Positive Airway Pressure | Oral Appliance
Number analyzed (Participants) | 65 | 54
percentage of NMAP to daytime MAP | 86.6 (8.18) | 87.9 (6.72)
Statistical Analysis 1: Comparison: Positive Airway Pressure vs Oral Appliance; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.3895, GLMM

5. Secondary Outcome: Mean Absolute Flow-Mediated Vasodilatation of the Brachial Artery by Vascular Ultrasound
Description: Mean absolute flow-mediated vasodilatation (FMD) of the brachial artery (i.e., the mean change in brachial artery diameter [in millimeters] from baseline to the value that is obtained after the cuff deflation) as measured by vascular ultrasound (VU) at the 6-month visit
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Positive Airway Pressure | Oral Appliance
Number analyzed (Participants) | 67 | 55
mm | 0.009 (0.0165) | 0.012 (0.0196)
Statistical Analysis 1: Comparison: Positive Airway Pressure vs Oral Appliance; Using analysis of covariance (robust MM regression), the outcome was regressed on an indicator variable for PAP vs. OA, baseline outcome, baseline apnea-hypopnea index, gender, site, baseline brachial-artery diameter, body mass index, age, and the interaction of gender and study arm. The latter allows for the possibility that treatment effect may differ between males and females. A Wald statistic was constructed for hypothesis testing; Test type: Superiority or Other; p = 0.3449, see Comments; Analysis of covariance with robust MM regression due to extreme residuals from initial fit showing strong departure from normal distribution

6. Secondary Outcome: Mean Relative Flow-Mediated Vasodilatation of the Brachial Artery by Vascular Ultrasound
Description: Mean relative flow-mediated vasodilatation (FMD) of the brachial artery (i.e., the mean change in brachial artery diameter from baseline to the value that is obtained after the cuff deflation, divided by the baseline value and multiplied by 100) as measured by vascular ultrasound (VU) at the 6-month visit
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Positive Airway Pressure | Oral Appliance
Number analyzed (Participants) | 67 | 55
percent change | 2.63 (4.550) | 3.51 (5.637)
Statistical Analysis 1: Comparison: Positive Airway Pressure vs Oral Appliance; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.1531, see Comments; [statistical method as in outcome 5, analysis 1]

ADVERSE EVENTS:
Time Frame: 6 months per patient
Description: Standardized questionnaire at each visit
Arm/Group | Positive Airway Pressure | Oral Appliance
Serious Adverse Events (participants affected / at risk) | 6/72 | 0/59
Other Adverse Events (participants affected / at risk) | 26/72 | 35/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Positive Airway Pressure (N=72) | Oral Appliance (N=59)
Non-ST elevated myocardial infarction (NSTEMI) (Cardiac disorders) | 1 | 0
Death-Acute Ischemic Stroke-Right Hemispheric Infarct (Nervous system disorders) | 1 | 0
Acute Hemorrhagic Stroke (Intraventricular Hemorrhage) (Nervous system disorders) | 1 | 0
Surgeries for Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 — Breast cancer surgery and separate surgery and hospital admission for catheter port placement for chemotherapy
Hyserectomy (Reproductive system and breast disorders) | 1 | 0
Dizziness (General disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Positive Airway Pressure (N=72) | Oral Appliance (N=59)
Motor Vehicle Accident (General disorders) | 1 | 1
Injury/Pain in Extremities (Musculoskeletal and connective tissue disorders) | 3 | 8
Hemodialysis catheter dislodgement (Blood and lymphatic system disorders) | 0 | 1
Cardiac Arrhythmia (Cardiac disorders) | 0 | 2
Sinusitis (Infections and infestations) | 1 | 2
Benign Skin Cyst Removal (Skin and subcutaneous tissue disorders) | 0 | 1
Tooth/Jaw Pain (Musculoskeletal and connective tissue disorders) | 0 | 4
Headache/Migraine (Nervous system disorders) | 1 | 1
Upper Respiratory Infection/Discomfort (Infections and infestations) | 3 | 10
Tooth Extraction (Infections and infestations) | 0 | 1
Spondylosis/Back Pain (Nervous system disorders) | 0 | 3
Ear Infection (Ear and labyrinth disorders) | 0 | 1
Worsened Depression (Psychiatric disorders) | 2 | 0
Abdominal Pain/Gastroenteritis (Gastrointestinal disorders) | 4 | 0
Cataract Surgery (Eye disorders) | 1 | 0
Esophageal Reflux (Gastrointestinal disorders) | 1 | 0
Increased High Blood Pressure (Cardiac disorders) | 4 | 0
Basal Cell Carcinoma Surgery (Skin and subcutaneous tissue disorders) | 1 | 0
Nasal Skin Irritation (Skin and subcutaneous tissue disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes